CLINICAL TRIAL: NCT02145000
Title: Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial to Assess the Efficacy and Safety of a Pentavalent Rotavirus Vaccine (BRV-PV) Against Severe Rotavirus Gastroenteritis Among Infants in Niger
Brief Title: Efficacy and Safety of a Pentavalent Rotavirus Vaccine (BRV-PV) Against Severe Rotavirus Gastroenteritis in Niger
Acronym: ROSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other); Serum Institute of India Pvt. Ltd. (Industry); FORSANI (Forum Santé Niger) (Unknown); Ministère de la Santé Publique, Niger (Unknown); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R822388
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Severe Rotavirus Gastroenteritis
Keywords: Rotavirus; Gastroenteritis; Diarrhea; Vaccine; Niger
MeSH Terms: conditions — Gastroenteritis; Diarrhea | interventions — Rotavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rotavirus vaccine (BRV-PV) (Experimental): Live attenuated bovine-human [UK] reassortant rotavirus vaccine manufactured by the Serum Institute of India, Limited (SIIL). The pentavalent vaccine (BRV-PV) contains rotavirus serotypes G1, G2, G3, G4, and G9 (≥5.6 log10 FFU/serotype/dose). The vaccine is in lyophilized form and supplied with 2.5 ml of citrate bicarbonate buffer that is added for reconstitution just before oral administration.
  Interventions: Biological: Rotavirus vaccine (BRV-PV)
- Placebo (Placebo Comparator): Same constituents as the active vaccine but without the viral antigens; manufactured by SIIL.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rotavirus vaccine (BRV-PV) — Three doses of BRV-PV containing ≥ Log10 5.6 FFU/Dose of each serotype G1, G2, G3, G4 and G9, or placebo, will be administered at 4 week intervals between doses (with a window of -1 to +4 weeks). The first administration will occur at 6-8 weeks of age.
  Arms: Rotavirus vaccine (BRV-PV)
Biological: Placebo
  Arms: Placebo

SUMMARY:
The study is a double-blinded, randomized, placebo-controlled, trial with two groups of infants receiving vaccine or placebo to assess the efficacy and safety of BRV-PV. Three doses of BRV-PV containing ≥ Log10 5.6 FFU/Dose of each serotype G1, G2, G3, G4 and G9 will be administered at 4 week intervals between doses. The first administration will occur at 6-8 weeks of age.

We hypothesize a difference in vaccine efficacy of three doses of BRV-PV vaccine vs. placebo against severe rotavirus gastroenteritis in healthy infants in Niger.

Active surveillance for gastroenteritis episodes will be conducted throughout the trial. Surveillance for adverse events will be carried out among all children from the time of first vaccination and 28 days post-Dose 3. Surveillance for all serious adverse events, including intussusception and death, will be conducted on all participants until they each reach two years of age.

To assess the effect of prenatal nutrition supplementation on infant immune response to the BRV-PV vaccine, study villages in the immunogenicity sub-cohort will be randomized in a 1:1:1 ratio to provide pregnant women with daily iron-folate, multiple micronutrients or a lipid-based nutrition supplement. Infants of participating women, if eligible at 6-8 weeks of age, will be randomized in a 1:1 ratio to receive three doses of vaccine or placebo and enter the main trial as part of the immunogenicity sub-cohort.

ELIGIBILITY:
Inclusion Criteria:

1. aged 6-8 weeks at the time of inclusion
2. able to swallow and no history of vomiting within 24 hours
3. resident in Madarounfa Health District and within the catchment area of the central health facility
4. intending to remain in the study area for 2 years
5. parent/guardian providing written informed consent

Exclusion Criteria:

Any of the following will exclude an infant from randomization in the study:

1. known history of congenital abdominal disorders, intussusception, or abdominal surgery
2. receipt of intramuscular, oral, or intravenous corticosteroid treatment within 2 wks
3. receipt or planned administration of a blood transfusion or blood products, including immunoglobulins
4. any known immunodeficiency condition
5. any serious medical condition
6. any other condition in which, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or the parent/guardian's ability to give informed consent

Ages: 6 Weeks to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6586 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Laboratory-confirmed episode of severe rotavirus gastroenteritis | From 28 days post-Dose 3 until 117 cases are accrued or when all participating infants reach 2 years of age if 117 cases are not attained

SECONDARY OUTCOMES:
Laboratory-confirmed episode of rotavirus gastroenteritis of any severity | From 28 days post-Dose 3 to 1 year of age, from 1 to 2 years of age, and from 28 days post-Dose 3 to 2 years of age
Laboratory-confirmed episode of rotavirus gastroenteritis with a Vesikari score of ≥ 17 | From 28 days post-Dose 3 to 1 year of age, from 1 to 2 years of age, and from 28 days post-Dose 3 to 2 years of age
Laboratory-confirmed episode of severe rotavirus gastroenteritis due to rotavirus serotypes G1, G2, G3, G4 and G9 | From 28 days post-Dose 3 to 1 year of age, from 1 to 2 years of age, and from 28 days post-Dose 3 to 2 years of age
Episode of gastroenteritis of any cause | From 28 days post-Dose 3 to 1 year of age, from 1 to 2 years of age, and from 28 days post-Dose 3 to 2 years of age
Hospitalization due to laboratory-confirmed cases of rotavirus gastroenteritis of any cause | From 28 days post-Dose 3 to 1 year of age, from 1 to 2 years of age, and from 28 days post-Dose 3 to 2 years of age
Hospitalization of any cause | From 28 days post-Dose 3 to 1 year of age, from 1 to 2 years of age, and from 28 days post-Dose 3 to 2 years of age
Any adverse health event | From the time of Dose 1 to 28 days post-Dose 3
Serious adverse events | From the time of Dose 1 until 2 years of age
Anti-rotavirus IgA sero-response rate | 28 days post-Dose 3
Anti-rotavirus IgA geometric mean titres | 28 days post-Dose 3

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Isanaka, ScD, Principal Investigator — Epicentre; Rebecca Grais, PhD, Study Director — Epicentre
Locations (1):
- Madarounfa Health District, Madarounfa, Maradi Region, Niger

REFERENCES:
- [Derived] Sudfeld CR, Bliznashka L, Salifou A, Guindo O, Soumana I, Adehossi I, Langendorf C, Grais RF, Isanaka S. Evaluation of multiple micronutrient supplementation and medium-quantity lipid-based nutrient supplementation in pregnancy on child development in rural Niger: A secondary analysis of a cluster randomized controlled trial. PLoS Med. 2022 May 2;19(5):e1003984. doi: 10.1371/journal.pmed.1003984. eCollection 2022 May. PMID 35500028
- [Derived] Kohlmann K, Sudfeld CR, Garba S, Guindo O, Grais RF, Isanaka S. Exploring the relationships between wasting and stunting among a cohort of children under two years of age in Niger. BMC Public Health. 2021 Sep 21;21(1):1713. doi: 10.1186/s12889-021-11689-6. PMID 34548050
- [Derived] Isanaka S, Garba S, Plikaytis B, Malone McNeal M, Guindo O, Langendorf C, Adehossi E, Ciglenecki I, Grais RF. Immunogenicity of an oral rotavirus vaccine administered with prenatal nutritional support in Niger: A cluster randomized clinical trial. PLoS Med. 2021 Aug 10;18(8):e1003720. doi: 10.1371/journal.pmed.1003720. eCollection 2021 Aug. PMID 34375336
- [Derived] Isanaka S, Langendorf C, McNeal MM, Meyer N, Plikaytis B, Garba S, Sayinzoga-Makombe N, Soumana I, Guindo O, Makarimi R, Scherrer MF, Adehossi E, Ciglenecki I, Grais RF. Rotavirus vaccine efficacy up to 2 years of age and against diverse circulating rotavirus strains in Niger: Extended follow-up of a randomized controlled trial. PLoS Med. 2021 Jul 2;18(7):e1003655. doi: 10.1371/journal.pmed.1003655. eCollection 2021 Jul. PMID 34214095
- [Derived] Isanaka S, Kodish SR, Mamaty AA, Guindo O, Zeilani M, Grais RF. Acceptability and utilization of a lipid-based nutrient supplement formulated for pregnant women in rural Niger: a multi-methods study. BMC Nutr. 2019 Jul 1;5:34. doi: 10.1186/s40795-019-0298-3. eCollection 2019. PMID 32153947
- [Derived] Coldiron ME, Guindo O, Makarimi R, Soumana I, Matar Seck A, Garba S, Macher E, Isanaka S, Grais RF. Safety of a heat-stable rotavirus vaccine among children in Niger: Data from a phase 3, randomized, double-blind, placebo-controlled trial. Vaccine. 2018 Jun 14;36(25):3674-3680. doi: 10.1016/j.vaccine.2018.05.023. Epub 2018 May 8. PMID 29752026
- [Derived] Isanaka S, Guindo O, Langendorf C, Matar Seck A, Plikaytis BD, Sayinzoga-Makombe N, McNeal MM, Meyer N, Adehossi E, Djibo A, Jochum B, Grais RF. Efficacy of a Low-Cost, Heat-Stable Oral Rotavirus Vaccine in Niger. N Engl J Med. 2017 Mar 23;376(12):1121-1130. doi: 10.1056/NEJMoa1609462. PMID 28328346